CLINICAL TRIAL: NCT05773339
Title: Prognostic Value of AIMS65 Score to Predict Outcome in Patients With Acute Upper Gastrointestinal Bleeding
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Nessma Mahmoud Abbas, resident doctor at internal medecine department, Sohag University
Other Study IDs: Soh-Med-23-02-07
Record Dates: First submitted 2023-03-06; First posted 2023-03-17 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Patients With Acute Upper Gastrointestinal Bleeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: AIMS65 score — The AIMS65 score consists of five factors:
  (i)albumin (1 point for value less than 3.0 g/dL (30 g/L)). (ii)INR (1 point for value greater than 1.5) . (iii)altered mental status (1 point given if Glasgow coma score was less than 14 or if disorientation, lethargy, stupor, or coma was seen) (iv)systolic blood pressure (1 point for value less than 90 mmHg). (v)age (1 point for value greater than 65 years).

SUMMARY:
Prognostic Value of AIMS65 Score to predict outcome in patients with acute upper gastrointestinal bleeding

DETAILED DESCRIPTION:
Gastrointestinal (GI) bleeding is one of the most important disease presentations in the emergency department. The course of the disease ranges from a self-limiting process to a life-threatening condition that requires emergency intervention. Evaluation of severity and the need for endoscopic hemostasis are matters of immediate decision. several prognostic scoring systems have been used to predict outcomes of upper GI bleeding ,such as the Rockall score, Glasgow-Blatchford score (GBS), and the AIMS65 score, among which AIMS65 is relatively easy to remember and simple to calculate by using parameters routinely available in the ED and importantly does not require endoscopic variables for calculation..

The AIMS65 score consists of five factors:

(i)albumin (1 point for value less than 3.0 g/dL (30 g/L)). (ii)INR (1 point for value greater than 1.5) . (iii)altered mental status (1 point given if Glasgow coma score was less than 14 or if disorientation, lethargy, stupor, or coma was seen) (iv)systolic blood pressure (1 point for value less than 90 mmHg). (v)age (1 point for value greater than 65 years). AIMS65 score >1: high risk patients. AIMS65 score >2: consider ICU management and an urgent endoscopy following adequate volume resuscitation, while AIMS65 score of 0 can be considered for outpatient management.

AIMS65 score is a simple non-endoscopic risk score that can be applied in patients of acute upper gastrointestinal bleeding to risk stratify and to predict in-patient mortality, the need for blood transfusion, endoscopic therapy or ICU admission.

In a comparative study of AIMS65 score and GBS ,they found that the AIMS65 score was superior in predicting inpatient mortality from UGIB, while the GBS was superior for predicting the need for blood transfusion. Both scores were similar in predicting the composite clinical endpoint .

ELIGIBILITY:
Inclusion Criteria:

* o Patients above 18 years of age.

  * Patients with acute UGIB presenting within 24 hours of hemorrhage onset.
  * Endoscopic evaluation done after hospital admission.

Exclusion Criteria:

* o Patients denying for consent.

  * Patients with late presentation (>24 hours) after UGIB onset.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients above 18 years of age.
  * Patients with acute UGIB presenting within 24 hours of hemorrhage onset.
  * Endoscopic evaluation done after hospital admission.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
to evaluate the prognostic value of AIMS65 score in patients with upper gastrointestinal tract bleeding admitted to Sohag University Hospital. | 6 months
  blood transfusion endoscopic therapy ICU admission Need of surgery, incidence of rebleeding duration of hospital and ICU stay.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Saltzman JR, Tabak YP, Hyett BH, Sun X, Travis AC, Johannes RS. A simple risk score accurately predicts in-hospital mortality, length of stay, and cost in acute upper GI bleeding. Gastrointest Endosc. 2011 Dec;74(6):1215-24. doi: 10.1016/j.gie.2011.06.024. Epub 2011 Sep 10. PMID 21907980
- [Background] Bryant RV, Kuo P, Williamson K, Yam C, Schoeman MN, Holloway RH, Nguyen NQ. Performance of the Glasgow-Blatchford score in predicting clinical outcomes and intervention in hospitalized patients with upper GI bleeding. Gastrointest Endosc. 2013 Oct;78(4):576-83. doi: 10.1016/j.gie.2013.05.003. Epub 2013 Jun 18. PMID 23790755
- [Background] Thandassery RB, Sharma M, John AK, Al-Ejji KM, Wani H, Sultan K, Al-Mohannadi M, Yakoob R, Derbala M, Al-Dweik N, Butt MT, Al-Kaabi SR. Clinical Application of AIMS65 Scores to Predict Outcomes in Patients with Upper Gastrointestinal Hemorrhage. Clin Endosc. 2015 Sep;48(5):380-4. doi: 10.5946/ce.2015.48.5.380. Epub 2015 Sep 30. PMID 26473120
- [Background] Stanley AJ, Laine L, Dalton HR, Ngu JH, Schultz M, Abazi R, Zakko L, Thornton S, Wilkinson K, Khor CJ, Murray IA, Laursen SB; International Gastrointestinal Bleeding Consortium. Comparison of risk scoring systems for patients presenting with upper gastrointestinal bleeding: international multicentre prospective study. BMJ. 2017 Jan 4;356:i6432. doi: 10.1136/bmj.i6432. PMID 28053181